CLINICAL TRIAL: NCT06667895
Title: Influences of the Autonomic Nervous System on Experimental Pain Sensitization
Brief Title: Pain Perception and the Autonomic Nervous System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schweinhardt Petra (Other)
Responsible Party: Sponsor-Investigator, Schweinhardt Petra, Prof. Dr. med., Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: taVNS
Record Dates: First submitted 2024-09-06; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Autonomic Nervous System Modulation; Pain Perception; Pain Sensitivity; Central Sensitization; Vagus Nerve Stimulations

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two phases, a pilot phase and a main experimental phase. The two phases involve different outcome measures. Both phases follow a double-blinded, randomized, within-subject design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS (Experimental): Electrodes will be attached to the outer ear. Electrical stimulation pulses with a width of 250ms will be applied at a frequency of 25Hz. Stimulation intensity will be individually adjusted to be clearly perceived but not painful.
  Interventions: Other: respiratory gated taVNS; Other: random burst stimulation; Other: continuous stimulation
- Sham stimulation (Sham Comparator): Electrodes will be attached to the outer ear at a different position as for the taVNS. Electrical stimulation pulses with a width of 250ms will be applied at a frequency of 25Hz. Stimulation intensity will be individually adjusted to be clearly perceived but not painful.
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Other: respiratory gated taVNS — Electrical stimulation will be delivered in bursts during expiration
  Arms: taVNS
Other: random burst stimulation — Electrical stimulation will be delivered in bursts at random timepoints during the breathing cycle
  Arms: taVNS
Other: continuous stimulation — Electrical stimulation will be delivered continuously for 30sec followed by a 30sec break.
  Arms: taVNS
Other: Sham stimulation — Electrical stimulation will be identical to the taVNS, but the electrodes will be placed at a different position on the ear
  Arms: Sham stimulation

SUMMARY:
In this study, we want to investigate how pain processing and sensation are related to a certain part of the nervous system, the so-called autonomic nervous system.

For this purpose, we apply heat and pressure stimuli to the skin and test pain processing by means of ratings scales and sensory tests. Breathing, heart rate and sweat response are also measured. To assess the spinal cord level, we measure muscle response (measured by electromyography, EMG) to electrical stimulation. Additionally, sensory nerves will be stimulated at the ear and participants will also be given various questionnaires to complete.

DETAILED DESCRIPTION:
This study investigates the effects of autonomic regulation on pain perception and experimentally induced pain sensitivity. Participants come for one or two study visits, that will last approximately 3 hours. The study is divided into two phases: the pilot phase and the main experimental phase.

During the pilot phase, the perception of pressure and heat stimuli, as well as spinal excitability, will be assessed before and during different types of electrical stimulation of sensory nerves at the outer ear.

During the main experimental phase, skin sensitivity and spinal excitability will be assessed before and after repetitive heat stimulation and stimulation of sensory nerves at the outer ear.

In both study phases, the activity of the autonomic nervous system will be assessed throughout the experiment, and questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 and below 40 years of age
2. Good general health
3. Able to give informed consent

Exclusion Criteria:

1. Any major medical or psychiatric condition (e.g. heart disease, diabetes, autoimmune disorders, infectious diseases, major depressive disorder), any chronic pain condition, any respiratory problems, any acute pain at time of study
2. Inability to follow study instructions, e.g. due to language problems
3. Pregnancy (female participants will be asked if pregnancy could be possible)
4. Increased alcohol (>2 (for women)/4 (for men) standard glasses per day or >5 (for women)/4 (for men) glasses at least once a month within a few hours) or caffeine consumption (≥ 400mg per day)
5. Consumption of alcohol, drugs, analgesics within the last 24 h
6. Consumption of more than 100 mg of caffeine within the last 8 h
7. Scar tissue or generally reduced sensitivity in the designated testing site areas
8. Shoe size < 38 (if experiment is conducted at the feet)
9. History of cardiovascular disease or carotid artery disease
10. Medication or Substances inferring with the autonomic nervous system or with pain sensitivity (e.g. Benzodiazepines, Nicotine)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the Nociceptive Withdrawl Reflex | Before, during, and/or immediately after the intervention
  Muscle responses of the biceps fermoris to an electrical stimulation of the sural nerve will be measured using an electromyogramm

OTHER OUTCOMES:
Area of Secondary Hyperalgesia | Before and 20 min after the intervention
  Von Frey filaments will be used to assess the spatial extent of experimentally induced hyperalgesia
Changes of Pressure Pain Threshold | Before, during, and/or immediately after the intervention
  Pressure will be applied over the thenar eminance of the hand until the participant reports a painful sensation
Perceived Pain Intensity and Unpleasantness | Before, during, and/or immediately after the intervention
  Perceived intensity and unpleasantness of heat stimuli will be assessed using rating scales. The intensity rating scale ranges from 0, indicating no perception, to 100, indicating the pain threshold, and up to 200, indicating the most tolerable pain. The unpleasantness rating scale ranges from -100 for 'extremely unpleasant,' through 0 for 'neutral,' to 100 for 'extremely pleasant.
Change in Autonomic Nervous System Activity | Before, during, and up to 2 min after the intervention.
  The activity of the autonomic nervous system will be measures using electrocardiogramm and galvanic skin response

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, PhD, M Chiro Med, Principal Investigator — Balgrist University Hospital, University of Zurich, Zurich, Switzerland
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data of participants who gave informed consent for further use of their anonymized data will be made available upon request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The PID, the study protocol and the analytical code will be available after publication for a maximum duration of 10 years
Access Criteria: PID will be made available for research purposes only. Anonymized data of all outcome measures can be made available upon request to the sponsor-investigator.